CLINICAL TRIAL: NCT05195905
Title: Evaluation of Spinal Cord Ischemia and Mortality and Morbidity After Endovascular Repair of Pararenal and Thoracoabdominal Aortic Aneurysm Using Surgeon-Modified Endografts
Brief Title: PMEG for Repair of Pararenal and Thoracoabdominal Aortic Aneurysm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konstantinos Dean Arnaoutakis, MD (Other)
Responsible Party: Sponsor-Investigator, Konstantinos Dean Arnaoutakis, MD, Assistant Professor of Surgery, University of South Florida
Organization: University of South Florida (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY002613
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Pararenal Aortic Aneurysm; Thoracoabdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Physician-modified endografts (Experimental): For this clinical protocol, endografts which are commercially available will be modified in a sterile fashion on a back-table in the operating room.
  Interventions: Device: PMEG

INTERVENTIONS:
Device: PMEG — All devices that will be modified in this study protocol are commercially available in the United States. The commercially available endografts will be used to construct a fenestrated/branched device for this intervention.

SUMMARY:
The primary objective is to evaluate the safety and effectiveness of surgeon modified endografts for the treatment of pararenal and thoracoabdominal aortic pathology in patients who are not candidate for traditional open repair due to comorbid issues and their anatomy is not amenable to commercially available endografts.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Male or female, aged ≥18 years
3. Expected survival beyond 1 year following successful aneurysm repair
4. Anatomy that would require coverage of the celiac artery, superior mesenteric artery (SMA), and/or renal arteries if conventional, FDA-approved endograft were implanted to obtain adequate sealing zone length
5. Aneurysm of the thoracoabdominal or pararenal aorta with or without chronic dissection
6. Adequate proximal zone of fixation
7. Adequate distal zone of fixation
8. No more than 5 non-aneurysmal visceral (celiac, SMA, or renal) arteries with diameters between 4-12mm
9. Adequate arterial access for delivery system; use of iliac conduit is permitted as necessary

Exclusion Criteria:

1. Moderate-to-severe aortic neck calcification, thrombus, or tortuosity
2. Severe iliac stenosis, calcification, or tortuosity with no ability to perform a conduit
3. Proximal landing within zone 0 or 1
4. Inability to maintain at least one patent hypogastric artery
5. Freely ruptured aneurysm with hemodynamic instability
6. Non-ambulatory status
7. Severe CHF
8. Baseline eGFR < 30ml/min, unless currently on or to be initiating dialysis
9. Unstable angina
10. Stroke or MI within 3 months of planned treatment date
11. Active systemic infection and/or mycotic aneurysm
12. Uncorrectable coagulopathy or other bleeding diathesis
13. Known allergy to device material or contrast material that cannot be adequately pre-medicated
14. Body habitus that would preclude adequate fluoroscopic visualization of aorta
15. Pregnancy or lactation (confirmed per standard of care surgical practice)
16. Major, unrelated surgical procedure planned ≤30 days from endovascular repair
17. Patient is ≤30 days beyond primary endpoint for another investigative clinical drug/device trial
18. Social or psychological issues that would interfere with ability to comply with all study procedures for the duration of the study
19. Can be treated in accordance with the instructions for use with a legally marketed endovascular device, including a manufacturer-fabricated custom device
20. Can enroll in a manufacturer-sponsored clinical study at our institution or is willing and eligible to participate in a study with a manufacturer-made device at another institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with 30-day major adverse events from primary procedure | Day 30
  Major adverse events include: aortic-related mortality, major stroke, myocardial Infarction, permanent spinal cord ischemia, renal failure, bowel Ischemia (requiring laparotomy/bowel resection), respiratory failure (mechanical ventilation >72 hours or requiring tracheostomy), lower extremity ischemia, blood loss ≥1,000cc
Number of subjects with treatment success | Month 12
  Treatment success is defined as a composite of: technical success, device integrity (freedom from stent fractures), freedom from aortic enlargement ≥5mm compared to preoperative CT imaging, freedom from aortic rupture, freedom from reintervention for type I or III endoleak or patency-related event, freedom from conversion to open aneurysm repair, freedom from aneurysm-related mortality.

SECONDARY OUTCOMES:
Number of subjects with mortality, major adverse events, spinal cord ischemia | Day 30, Month 6, Month 12, Month 24, Month 36, Month 48, Month 60
  Mortality includes all-cause mortality. Major adverse events include: aortic-related mortality, major stroke, myocardial Infarction, permanent spinal cord ischemia, renal failure, bowel Ischemia (requiring laparotomy/bowel resection), respiratory failure (mechanical ventilation >72 hours or requiring tracheostomy), lower extremity ischemia, blood loss ≥1,000cc. Spinal cord ischemia data will include all incidence and degree of spinal cord ischemia.
Number of subjects with treatment success and freedom from secondary intervention | Day 30, Month 6, Month 12, Month 24, Month 36, Month 48, Month 60
  Treatment success is defined as a composite of: technical success, device integrity (freedom from stent fractures), freedom from aortic enlargement ≥5mm compared to preoperative CT imaging, freedom from aortic rupture, freedom from reintervention for type I or III endoleak or patency-related event, freedom from conversion to open aneurysm repair, freedom from aneurysm-related mortality. Freedom from secondary interventions includes interventions to treat malperfusion, rupture, aneurysm formation, aortic expansion, endoleak, device stenosis/occlusion, or access site complication.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Arnaoutakis, MD, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - Tampa General Hospital, Tampa, Florida
  - University of South Florida - South Tampa Campus, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dossabhoy SS, Simons JP, Flahive JM, Aiello FA, Sheth P, Arous EJ, Messina LM, Schanzer A. Fenestrated endovascular aortic aneurysm repair using physician-modified endovascular grafts versus company-manufactured devices. J Vasc Surg. 2018 Jun;67(6):1673-1683. doi: 10.1016/j.jvs.2017.10.055. Epub 2017 Dec 8. PMID 29224942
- [Background] Oderich GS, Ribeiro MS, Sandri GA, Tenorio ER, Hofer JM, Mendes BC, Chini J, Cha S. Evolution from physician-modified to company-manufactured fenestrated-branched endografts to treat pararenal and thoracoabdominal aortic aneurysms. J Vasc Surg. 2019 Jul;70(1):31-42.e7. doi: 10.1016/j.jvs.2018.09.063. Epub 2018 Dec 21. PMID 30583902
- [Background] Eagleton MJ, Follansbee M, Wolski K, Mastracci T, Kuramochi Y. Fenestrated and branched endovascular aneurysm repair outcomes for type II and III thoracoabdominal aortic aneurysms. J Vasc Surg. 2016 Apr;63(4):930-42. doi: 10.1016/j.jvs.2015.10.095. Epub 2016 Jan 11. PMID 26792544
- [Background] Schanzer A, Simons JP, Flahive J, Durgin J, Aiello FA, Doucet D, Steppacher R, Messina LM. Outcomes of fenestrated and branched endovascular repair of complex abdominal and thoracoabdominal aortic aneurysms. J Vasc Surg. 2017 Sep;66(3):687-694. doi: 10.1016/j.jvs.2016.12.111. Epub 2017 Mar 1. PMID 28259577
- [Background] Oderich GS, Ribeiro M, Hofer J, Wigham J, Cha S, Chini J, Macedo TA, Gloviczki P. Prospective, nonrandomized study to evaluate endovascular repair of pararenal and thoracoabdominal aortic aneurysms using fenestrated-branched endografts based on supraceliac sealing zones. J Vasc Surg. 2017 May;65(5):1249-1259.e10. doi: 10.1016/j.jvs.2016.09.038. Epub 2016 Dec 13. PMID 27986479
- [Background] Conrad MF, Crawford RS, Davison JK, Cambria RP. Thoracoabdominal aneurysm repair: a 20-year perspective. Ann Thorac Surg. 2007 Feb;83(2):S856-61; discussion S890-2. doi: 10.1016/j.athoracsur.2006.10.096. PMID 17257941
- [Background] Coselli JS, Bozinovski J, LeMaire SA. Open surgical repair of 2286 thoracoabdominal aortic aneurysms. Ann Thorac Surg. 2007 Feb;83(2):S862-4; discussion S890-2. doi: 10.1016/j.athoracsur.2006.10.088. PMID 17257942
- [Background] Schepens MA, Heijmen RH, Ranschaert W, Sonker U, Morshuis WJ. Thoracoabdominal aortic aneurysm repair: results of conventional open surgery. Eur J Vasc Endovasc Surg. 2009 Jun;37(6):640-5. doi: 10.1016/j.ejvs.2009.03.011. Epub 2009 Apr 11. PMID 19362499
- [Background] Arnaoutakis DJ, Scali ST, Beck AW, Kubilis P, Huber TS, Martin AJ, Laquian L, Back M, Giles KA, Fatima J, Beaver TM, Upchurch GR Jr. Comparative outcomes of open, hybrid, and fenestrated branched endovascular repair of extent II and III thoracoabdominal aortic aneurysms. J Vasc Surg. 2020 May;71(5):1503-1514. doi: 10.1016/j.jvs.2019.08.236. Epub 2019 Nov 11. PMID 31727462
- [Background] Scali ST, Kim M, Kubilis P, Feezor RJ, Giles KA, Miller B, Fatima J, Huber TS, Berceli SA, Back M, Beck AW. Implementation of a bundled protocol significantly reduces risk of spinal cord ischemia after branched or fenestrated endovascular aortic repair. J Vasc Surg. 2018 Feb;67(2):409-423.e4. doi: 10.1016/j.jvs.2017.05.136. Epub 2017 Oct 7. PMID 29017806